CLINICAL TRIAL: NCT00971490
Title: Effects of a 4-week Acu-Transcutaneous Electrical Nerve Stimulation (Acu-TENS) Program on Subjects With Stable Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Prof. Alice Jones, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CRE-2007.158-T
Record Dates: First submitted 2009-07-28; First posted 2009-09-03 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; FEV1; beta endorphin; SGRQ; Acu-TENS
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Group 1 (Experimental)
  Interventions: Device: Acu-TENS (Transcutaneous electrical nerve stimulation)
- Group 2 (Placebo Comparator)
  Interventions: Device: Acu-TENS (Transcutaneous electrical nerve stimulation)
- Group 3 (Sham Comparator)
  Interventions: Device: Acu-TENS (Transcutaneous electrical nerve stimulation)

INTERVENTIONS:
Device: Acu-TENS (Transcutaneous electrical nerve stimulation) — Transcutaneous electrical nerve stimulation applied onto acupuncture point
  Arms: Group 1
Device: Acu-TENS (Transcutaneous electrical nerve stimulation) — Similar to Group 1 but without electrical stimulation
  Arms: Group 2
Device: Acu-TENS (Transcutaneous electrical nerve stimulation) — Similar to Group 1 but applied onto non acupuncture point
  Arms: Group 3

SUMMARY:
The objectives of this study are to investigate the effectiveness of Acu-TENS (transcutaneous electrical nerve stimulation applied on acupoints) on lung functions and quality of life and to explore the associated underlying mechanisms in subjects with COPD.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis with COPD

Exclusion Criteria:

* allergic to gel
* unable to perform spirometry
* unable to communicate
* no history of infection or exacerbation of respiratory symptoms

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1), forced vital capacity (FVC) | measured before and after the 4-week program

SECONDARY OUTCOMES:
beta endorphin, St George Respiratory Questionnaire (SGRQ) | measured before and after the 4-week program

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong, China